CLINICAL TRIAL: NCT05713331
Title: Web-based Professional Development for School Mental Health Providers in Evidence-Based Practices for Attention and Behavior Challenges
Brief Title: Web-based Professional Development for SMHPs in Evidence-Based Practices for Attention and Behavior Challenges
Acronym: CLS-R
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: School closures during COVID-19 precluded study activities
Sponsor: University of California, San Francisco (Other)
Collaborators: Institute of Education Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R305A170338
Record Dates: First submitted 2022-10-31; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CLS-R (Experimental): Web-based remote training for school mental health providers
  Interventions: Behavioral: CLS-R
- CLS (Active Comparator): In-person training for school mental health providers
  Interventions: Behavioral: CLS-R

INTERVENTIONS:
Behavioral: CLS-R — CLS-R Training includes school provider training in CLS via web platform and videoconferencing for workshops, consultation and coaching.CLS is a 10-12 week program and includes school, parent, and student components which are integrated via joint teacher, parent, and student meetings and use of integrated behavioral programs in the classroom and home.

SUMMARY:
This study develops a web-based PD (CLS-R) to provide SSWs with remote training in EBPs for attention and behavior problems. CLS-R is designed to be usable, feasible, portable, accessible, and acceptable - ingredients which have been identified as necessary for the sustainability of school-based programs. The study evaluates the usability, feasibility, acceptability, fidelity of implementation, and preliminary effects on student outcomes.

DETAILED DESCRIPTION:
1. Title of Project: Web-Based Professional Development for School Mental Health Providers in Evidence-Based Practices for Attention and Behavior Challenges
2. RFA Topic and Goal: Social and Behavioral Context for Academic Learning, Goal 2
3. Purpose: Development of a web-based professional development program (PD) for school mental health providers to gain the skills needed to implement evidence-based practices (EBPs) for attention and behavior problems.
4. Setting: The research will be conducted in elementary schools within San Francisco Unified School District (SFUSD).
5. Sample: Participants will include SFUSD school social workers (SSWs), students, parents and teachers.
6. Professional Development to be developed: The Collaborative Life Skills (CLS) program will be developed into a web-based format (CLS-R) with all training and consultation provided remotely via videoconferencing. Includes EBP skill modules for consulting with teachers and parents and working with students directly.
7. Control Condition: N/A
8. Research design and methods: (1)Open Trials and Refinement: CLS-R will be field tested with 4 SSWs delivering the intervention to students, parents, and teachers. Modification and refinement of materials, manuals, and procedures will follow each trial based on questionnaire data and focus groups. Outcomes will evaluate usability, feasability, and acceptability, implementation fidelity, preliminary effects on student outcomes, and post-training sustainability of SSW EBP skill use. (2) Pilot Study: Using a randomized design, we will compare CLS-R and CLS. Six SSWs will receive CLS-R and 6 SSWs will receive CLS. To temporarily conduct study during COVID-19 school closures, we will test feasbility, usability and accesptability of the fully remote CLS parent component.
9. Key measures: Measures of process (training fidelity, attendance), feasibility, usability, and acceptability will be obtained.
10. Data analytic strategy: CLS-R usability and feasibility will focus on qualitative analysis of themes from focus groups, quantitative analyses of rating scales, and descriptive analyses of functionality.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 7-11, 2nd-5th grades
* Presence of academic and social problems related to inattention and/or hyperactivity/impulsivity (as judged by school SSW)
* Six or more inattention symptoms and/or six or more hyperactive/impulsive symptoms endorsed across parent and teacher rating scales (using an either-or algorithm, such that a symptom is counted as being present if either parent or teacher endorses it as occurring 'often' or 'very often')
* Functional impairment reported by either parent or teacher on the IRS (score of 3 or greater)
* Caretaker available and consents to participate in treatment
* Currently attending a participating school full-time

Exclusion Criteria:

* Presence of conditions that are incompatible with this study's treatment:

  * severe visual or hearing impairment,
  * severe language delay,
  * psychosis,
  * pervasive developmental disorder
  * Parent or child does not read or speak English or does not read or speak Spanish for our Spanish language implementation of CLS (inability to complete assessment measures or participate in group treatments).
* Child is in an all-day special education classroom (children in these classrooms are frequently receiving intensive behavior modification programs such that the intervention would be expected to require modification for use in these settings)
* Children taking psychotropic medication for any reason other than to treat ADHD
* Children planning to change (start or stop) psychotropic medication
* Children who have changed a regimen of psychotropic medication (started or stopped) within 30 days prior to screening

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 79 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Symptoms of Attention Deficit Hyperactivity Disorder as defined by DSMV | Change from baseline to post-treatment
  Parent and teacher rating scale

SECONDARY OUTCOMES:
Homework Problems Checklist (HPC) | Change from baseline to post-treatment
  Parent-rated scale
Children's Organizational Skills Scale (COSS) | Change from baseline to post-treatment
  Parent and teacher rating scale
Symptoms of Oppositional Defiant Disorder as defined by DSMV | Change from baseline to post-treatment
  Parent and teacher rating scale
Strengths and Difficulties Questionnaire | Change from baseline to post-treatment
  Parent and teacher rating scale
Clinical Global Improvement | Change from baseline to post-treatment
  Parent and teacher rating scale
School Mental Health Provider Rating of Skill Competence, Motivation and Knowledge | Change from baseline to post-treatment
  School mental health provider rating scale
Alabama Parenting Questionnaire | Change from baseline to post-treatment
  Parent rating scale
Parenting Stress Index | Change from baseline to post-treatment
  Parent rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Linda Pfiffner, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - HALP Clinic, Children's Center at Langley Porter, UCSF, San Francisco, California
  - University of California San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No